CLINICAL TRIAL: NCT07381322
Title: A Study on the Accurate Evaluation of Pseudoprogression of Rectal Cancer Immunotherapy Based on Multitemporal and Multiparameter MRI
Status: Recruiting | Type: Observational
Sponsor: Peiyi Xie (Other)
Collaborators: Xinyi City People's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Peiyi Xie, associate chief physician, Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Other Study IDs: 2026ZSLYEC-028
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one group: one group

SUMMARY:
This project aims to use multi-temporal, multi-parameter MRI features, blood biomarkers, and clinical indicators to accurately assess pseudoprogression following immunotherapy in rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Rectal cancer confirmed by biopsy pathology;
2. Clinical stage II-IV determined by imaging examinations;
3. Decided by the MDT team to receive immunotherapy (monotherapy with PD-1/PD-L1 inhibitors or in combination with CTLA-4 inhibitors), without prior treatment of any other kind;
4. Multiparametric MRI images of the rectum obtained within 2 weeks before immunotherapy, and at 6 and 12 weeks after treatment;
5. Follow-up CT/MRI data available; evaluation conducted according to the iRECEST criteria, or surgical resection performed to obtain postoperative pathological results, which are necessary for assessing the efficacy of immunotherapy and diagnosing pseudoprogression versus true progression;
6. Blood test parameters (IL-8, NLR, LDH, S100) and clinical indicators (KPS score, CEA level, T-stage) measured within 2 weeks before immunotherapy, and at 6 and 12 weeks after treatment;
7. In cases where imaging suggests disease progression, pathological biopsy or surgical pathology results must be available.
8. The overall survival period is more than 3 months, and the patient does not have any other uncontrollable diseases;
9. The patient has been fully informed and has signed the informed consent form.

Exclusion Criteria:

1. The primary tumor lesion has been surgically removed at the time of initial diagnosis;
2. History of other malignant tumors;
3. Unable to sign informed consent or complete the trial due to physical or psychological illness;
4. Pregnant or lactating women;
5. Those who are allergic to gadolinium-containing contrast agents or contraindicated to undergo enhanced MRI examination, or those who are claustrophobic or have other contraindications to MRI examination and cannot undergo MRI examination;
6. History of autoimmune diseases such as inflammatory bowel disease;
7. Treatment interruption due to serious complications related to immunotherapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rectal cancer treaded with immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The area under curve (AUC) of receive operating characteristic (ROC) curves of models in prediction pseudoprogression after rectal cancer immunotherapy | From date of baseline MRI to date of preoperative MRI

SECONDARY OUTCOMES:
The specificity of models in prediction pseudoprogression | From date of baseline MRI to date of preoperative MRI
The sensitivity of models in prediction pseudoprogression | From date of baseline MRI to date of preoperative MRI
The positive predictive value of models in prediction pseudoprogression | From date of baseline MRI to date of preoperative MRI
The negative predictive value of models in prediction pseudoprogression | From date of baseline MRI to date of preoperative MRI
The accuracy of models in prediction pseudoprogression | From date of baseline MRI to date of preoperative MRI
Disease-free survival and overall survival | From date of enrollement until the date of first documented progression or date of death from any cause,whichever came first,assessed up to 60 months
patients are divided into: iCPD patients are classified as the 'tumor progression group after immunotherapy,' while iCR, iPR, and iSD patients are classified as the 'non-tumor progression group after immunotherapy. | From date of enrollement until the date of first documented progression or date of death from any cause,whichever came first,assessed up to 60 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sixth affiliated hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Xinyi People's hospital, Maoming, Guangdong